CLINICAL TRIAL: NCT03222375
Title: The Home-Use of Semiconducting QUantum Excitonic Device: Image Converter/Sound Converter/Electromagnetic Converter to Improve Communicative Efforts, Speech, Language and Related Cognitive Functions in Children With Autism
Brief Title: SQUED™ Series 28.1 Home-use and Treatment of Autowave Reverberator of Autism
Acronym: SQUED™
Status: Recruiting | Type: Observational
Sponsor: American Federation of Medical Synergetics (Other)
Collaborators: Clinic of Synergetics, Department of Neurology/Neuropsychology WOMS (Unknown); Institute of Medical Synergetics, Department of Cognitive Neurology WOMS (Unknown); Laboratory of Neurocomputational Active Media WOMS (Unknown); SQUED, Inc., USA (Unknown); Center of Synergetics, Universität Stuttgart, Germany (Unknown); Ivan Franko National University of Lviv, Ukraine (Unknown); Danylo Halytsky Lviv National Medical University (Other); World Organization of Medical Synergetics (Other); World Autism Center, American Federation of Medical Synergetics (Unknown)
Responsible Party: Sponsor
Other Study IDs: SQUED™ series 28.1 home-use
Record Dates: First submitted 2017-07-13; First posted 2017-07-19 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Neurodevelopmental Disorders; Mental Disorders; Asperger's Syndrome; Neurobehavioral Manifestations; Nervous System Diseases
Keywords: Yaroshuk's MEGA-DISCOVERY · DIAGNOSTICS · TREATMENT; Yaroshuk's Scientific Medical School; Center of Synergetics; Controlling spatiotemporal chaos/Dr. Synergetic; Autowave processes in Medicine; Autowave Reverberator; Bifurcation of Dynamic systems on a plane; Spiral Autowaves; Drift of Spiral Autowaves; Excitable medium and Cellular Automata; Stochastic Resonance and Coherence Resonance; Autowaves/SQUED; Theory of Semiconducting QUantum Excitonic Device
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Neurodevelopmental Disorders; Mental Disorders; Asperger Syndrome; Neurobehavioral Manifestations; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Autism: Individuals with autism will have either Image converter (iSQUED™) for Hysteresis of Spiral Autowaves, Sound converter (sSQUED™) for Drift of Spiral Autowaves or Electromagnetic converter (eSQUED™) for Annihilation Autowave reverberator.
  Interventions: Device: SQUED™ series 28.1 home-use

INTERVENTIONS:
Device: SQUED™ series 28.1 home-use — Semiconducting QUantum Excitonic Device - artifificial active medium, where the processes of self-organization lead to creation and converter of Autowaves energy.
  Some autowaves have the properties of quasi-particles!

SUMMARY:
Locomotor, transport and information functions in human body systems are carried out by active media in autowave regimes! Any living organism is a (micro-macro-mega) hierarchy of autowave subsystems-an ensemble of loosely coupled subsystems of a simpler structure. From the highest levels of the hierarchy, Autowave Codes-Signals arrive, which determine the transitions of subsystems from one autowave regime to another Autowave interaction (of Complex Coherent Action). Autowave interaction is a process associated with the evolution and interaction of spatial and wave structures in the active media of the organism.

Chaos in organism functioning tells about health. Periodicity - Autowave reverberator may presage a disease - Autism Spectrum Disorder; Chaotic nature of oscillations in active media of physiological systems is more optimal for their vital functions than periodic one. Firstly, systems that function in chaotic regimes, can re-arrange themselves faster and easier in case of change of environmental conditions, i.e. the so called adaptive control is more easily implemented in them. Secondly, "spreading" of oscillations strength along comparatively wide frequency band takes place in chaotic regime.

When an organism is young and healthy, physiological systems show the elements of chaotic behavior, i.e. irregularity and chaotic dynamics are the extremely important characteristics of health. Decrease in changeability and appearance of stable periodicity of Autowave reverberator are often connected with Autism.

The main purpose is to study brain plasticity (the changes that occur in the brain through Autowave reverberator) in children with autism. Research suggests that during development, the brains of children may change in response to their Autowave reverberator differently than the brains of typically developing individuals. Investigators want to understand why and how this difference may contribute to the symptoms of autism spectrum disorder (ASD). In this study, the investigators will be examining the effects of non-invasive neuromodulation SQUED™ series 28.1 home-use for Treatment of Autowave reverberator of Autism.

Integrative Team World Organization of Medical Synergetics (WOMS) - collaborations between physicians and researchers with expertise in biostatistics, physics, mathematics, engineering, and computer science.

DETAILED DESCRIPTION:
Autowave Reverberator:

1. Proved that, a Autowave Reverberator appears a result of a rupture of Autowave front; initial conditions - Natal Trauma:

   1.1 Proved that, such a rupture may occur, via collision of the Autowave front with a nonexcitable obstacle - brain injury or injury of vertebral;

   1.2 Proved that, such a rupture may occur by loss of excitation in a certain region of the Active medium - cerebral anoxia;

   1.3 Locomotor, Transport and Information functions in the physiological systems, and Communicative Efforts, Speech, Language and Related Cognitive Functions this is Autowave processes in Active media.
2. An important feature of reverberators is that these Autowave sources have the highest frequency. By generating pulses at a maximum frequency such sources force out self-pacemakers of any other types from the medium. As a result, the Active medium is filled with only Spiral Autowaves:

   2.1 The basic parameters of a reverberator are the frequency of generated waves, the critical dimension and characteristics of the structure of the kernel, and the velocity of the kernel in space, at Drift of Spiral Autowaves and/or Annihilation of Spiral Autowaves, or Multiplication of Spiral Autowaves;

   2.2 Commonly, there are two characteristic regions in a reverberator: a kernel having an excitation "tongue" entering it and Spiral Autowaves generated by the kernel - one spiral/two spirals/three spirals/four spirals; central filament of the Autowaves-branch rotates Left/Right;

   2.3 The kernel can have the form of a circle or a ring, a so-called "anomalous" kernel. If the source drifts, the form of the kernel is involved and can hardly be determined unambiguously.
3. Proved that, the reverberator is not tied to any structure in the Active medium:

   3.1 Proved that, due to this property, reverberators can Appear and Disappear in the different Endoderm/Mesoderm/Ectoderm of the Active media, and at different locations of the Active medium;

   3.2 Proved that, due to this property, reverberators can Appear and Disappear in the Ectodermal Active media - Brain/spinal cord/hair/Skin; central filament of the endogenous Brain branch/exogenous Skin-branch;

   3.3 Proved that, reverberators can Observe on the skin, Spiral Autowaves generated by the kernel - one spiral/two spirals/three spirals/four spirals; central filament of the Pileous-branch rotates Left/Right.
4. Proved, Center of Synergetics/Dr. Synergetic (the name of a new physician - Nonlinear Control of Autowaves chaos in Active media), Nonlinear Control of Autowaves reverberators:

   4.1 Proved, Nonlinear Control of Autowaves reverberators: Hysteresis of Spiral Autowaves, Drift of Spiral Autowaves and Annihilation of Spiral Autowaves.
5. Treatment of Autowave Reverberator of Autism (this will be administered by Presence of Clinical protocol CRF-SQUED™):

5.1 Diagnostics of Autowave reverberators and Mathematical Modeling of Autowave reverberators in Active media + Algorithmic approach;

5.2 Computational Simulation of Autowave reverberator and Mathematical Modeling of treatment code (Trade Secret) + creation Active medium SQUED™ for a patient;

5.3 Recording for a patient of treatment code (Trade Secret) on the Image Converter/Sound Converter/Electromagnetic Converter + Autowave regime: Hysteresis of Spiral Autowaves; Drift of Spiral Autowaves; Annihilation of Autowave reverberator;

5.4 SQUED™ Treatment of Autowave reverberator of Autism (Novel type energy/Non-invasive) + Semiconducting Quantum Excitonic Device - artificial active medium, where the processes of self-organization lead to creation and converter of Autowaves energy.

Some autowaves have the properties of quasi-particles!

Participants in the study will be asked to do the following things:

* Grant permission for the researchers to view medical/psychological and/or educational and/or speech records associated with the diagnosis of autism.
* Complete a questionnaire and provide a health history.
* Complete evaluations by our study team to assess the diagnosis and gain a clearer understanding of the participant's current functioning.
* Give to our study team of Photo of Autowave Reverberator - Presence on the Skin of the interruption of Autowave front (interruption of hair separatrix - dorsal/ventral) and/or Photo of Spiral Autowaves, generated by the kernel of Autowave Reverberator - the kernel having an excitation "tongue".
* Give to our study team of Graphics on tracing paper of Autowave Reverberator - Presence on the Skin of the interruption of Autowave front (interruption of hair separatrix - dorsal/ventral) and/or Graphics on tracing paper of Spiral Autowaves, generated by the kernel of Autowave Reverberator - the kernel having an excitation "tongue".
* Complete several tasks and training interventions that involve such things as learning new words or pictures, saying words out loud, or naming objects.
* Complete several tasks and training interventions that involve such things as creation pictures iSQUED™ and music compositions sSQUED™.
* Give permission to audio and video-tape test sessions for later scoring and observation.
* Give permission to audio or video-tape in the Home environment or classroom using non-intrusive audio-visual recording devices.
* Participate in computerized tasks of Image converter SQUED™ (iSQUED™). The software/device poses no risk and is non-invasive.
* Participate in computerized tasks of Sound converter SQUED™ (sSQUED™). The software/device poses no risk and is non-invasive.
* Participate in computerized tasks of Electromagnetic converter SQUED™ (eSQUED™). The device/software poses no risk and is non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism or related conditions.
* History of Late complications at Natal Trauma:

  1. Cerebral level of Natal Trauma - brain injury;
  2. Cervical level of Natal Trauma - injury of vertebral;
  3. Cerebral anoxia.
* Identified language deficit(s) and/or other cognitive or behavioral impairments (which will be specific to each sub-study).
* Adequate ability to perform the research tasks set for the Age level:

  1. Infant - greater than 1 month to 2 years of age;
  2. Child - greater than 2 to 12 years of age;
  3. Adolescent - greater than 12 through 21 years of age.
* Presence on the Skin of the interruption of Autowave front (interruption of hair separatrix - dorsal/ventral) and/or of the Autowave Reverberators:

  1. Photo of Spiral Autowaves, generated by the kernel of Autowave Reverberator - the kernel having an excitation "tongue";
  2. Graphics on tracing paper of Spiral Autowaves, generated by the kernel of Autowave Reverberator - the kernel having an excitation "tongue".
* Presence of Clinical protocol CRF-SQUED™:

  1. Diagnostics of Autowave reverberators and Nonlinear Control of Autowave reverberators in Active media (Autowave interaction of patient - Algorithmic approach);
  2. Mathematical Modeling of Autowave Reverberator and Computational Simulation of the treatment code (Trade Secret), and creation Active medium SQUED™ for a patient;
  3. Recording for a patient of treatment code (Trade Secret) - Autowave regime: Hysteresis of Spiral Autowaves; Drift of Spiral Autowaves; Annihilation of Autowave reverberator.
* Magnetogram of region of Home-use and Geographic coordinates of Home-use.

Exclusion Criteria:

* Peripheral blindness - precludes use of Image converter SQUED™ (iSQUED™).
* Peripheral deafness - precludes use of Sound converter SQUED™ (sSQUED™).
* Any implanted metal device - precludes use of Electromagnetic converter SQUED™ (eSQUED™).
* Any implanted cardiac pacemaker - precludes use of Electromagnetic converter SQUED™ (eSQUED™).

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be 1 month to 21 years of age, diagnosed with autism by independent clinicians and confirmed by formal assessment (e.g., CDI, ADOS, Bayley, Sensory Profile), and with receptive and expressive vocabulary levels of ≥ 3 years age-equivalent, as assessed by standardized measures. Additionally, the Autism Diagnostic Interview will be administered to caregivers in order to appropriately identify specific areas (regarding speech, language and cognition) in which participants are experiencing the most difficulty. The experimental group will consist of children (Infant, Child and Adolescent) with Autowave reverberators of Autism (n = 80): 1/2/3/4 armed/Left/Right_Spiral Autowaves.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
SQUED™ software of patient | Personal Autowave Diagnostics/Personal Autowave Therapy - through study completion, an average of 1 year
  This will be administered by Presence of Clinical protocol CRF-SQUED™and creation Active medium SQUED™ for a patient.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliya Yaroshuk, M.D.s. Ph.D., Principal Investigator — World Autism Center, American Federation of Medical Synergetics, Department of Neurology; Cognitive Neurology/Neuropsychology WOMS; Yuriy Fihol, M.D.s. Ph.D., Principal Investigator — Clinic of Synergetics, Department of Neurology; Cognitive Neurology/Neuropsychology of the World Organization of Medical Synergetics
Locations (2):
- World Autism Center, American Federation of Medical Synergetics, Department of Neurology; Cognitive Neurology/Neuropsychology WOMS, Louisville, Kentucky, United States
- Clinic of Synergetics, Department of Neurology; Cognitive Neurology/Neuropsychology of the World Organization of Medical Synergetics, Lviv, Solonka Village, Urozayna Street 41, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
This will be administered by Presence of Clinical protocol CRF-SQUED™ and creation Active medium SQUED™ of Patient.
Supporting Information: CSR
Time Frame: Personal Autowave Diagnostics/Personal Autowave Therapy
Access Criteria: SQUED™ software - Active medium SQUED™ of Patient

REFERENCES:
- See also: Center of Synergetics, Universität Stuttgart, Germany — http://itp1.uni-stuttgart.de/en/institut/arbeitsgruppen/haken/cos.php
- See also: Headquarters of World Organization of Medical Synergetics, Lviv - Solonka ( 49°45'56.6"N 23°59'53.7"E ) — http://www.google.com/maps/place/49%C2%B045'56.6%22N+23%C2%B059'53.7%22E/@49.7659965,23.9979761,690m/data=!3m1!1e3!4m5!3m4!1s0x0:0x0!8m2!3d49.7657222!4d23.99825
- See also: Yaroshuk's Scientific Medical School — http://plus.google.com/communities/101353132492658668565
- See also: Autowave processes in Medicine - book — http://www.springer.com/in/book/9789027723796
- See also: Nonlinear Control - book — https://www.amazon.com/Self-Organized-Biological-Dynamics-Nonlinear-Control/dp/0521026075
- See also: Drift of spiral wave in excitable media — http://www.scholarpedia.org/article/Drift_of_spiral_waves
- See also: Some classic types of reverberator evolution - Hysteresis width — http://cdn.intechopen.com/pdfs-wm/46160.pdf
- See also: Efficient control of spiral wave location in an excitable medium — http://iopscience.iop.org/article/10.1088/1367-2630/10/1/015003
- See also: Autowave reverberator — http://en.wikipedia.org/wiki/Autowave_reverberator
- See also: Modelling excitable media — https://en.wikipedia.org/wiki/Excitable_medium
- See also: Excitable media — http://www.scholarpedia.org/article/Excitable_media
- See also: Theory of bifurcations of dynamic systems on a plane - eBook "Mathematical on the Skin" — https://archive.org/details/nasa_techdoc_19710012507